CLINICAL TRIAL: NCT03051490
Title: A Phase 3, Randomized, Open-Label, Assessor-Blind, Non-Inferiority, Active-Comparator Study Evaluating the Efficacy and Safety of Liprotamase in Subjects With Cystic Fibrosis-Related Exocrine Pancreatic Insufficiency
Brief Title: RESULT: Reliable, Emergent Solution Using Liprotamase Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN-EPI3333
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-01

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — liprotamase lipase

STUDY DESIGN:
Masking Description: unblinded to treatment randomization; blinded to primary efficacy variable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liprotamase (Experimental): Individually-optimized dose to be administered orally
  Interventions: Drug: Liprotamase
- porcine PERT (Active Comparator): Individually-optimized dose to be administered orally
  Interventions: Drug: porcine PERT

INTERVENTIONS:
Drug: Liprotamase — oral, soluble, non-enterically coated, non-porcine, pancreatic enzyme replacement
  Arms: Liprotamase
Drug: porcine PERT — oral, enterically-coated, pig-derived, pancreatic enzyme replacement
  Arms: porcine PERT

SUMMARY:
Liprotamase powder is a non-porcine, soluble and stable mixture of biotechnology-derived lipase, protease, and amylase digestive enzymes. The purpose of the present study is to to evaluate the non-inferiority of liprotamase compared with porcine-derived, enterically-coated pancreatic enzyme replacement therapy (PERT). The primary efficacy endpoint of the study will be comparative efficacy measured as the change from baseline in the coefficient of fat absorption (CFA) in Cystic Fibrosis patients with exocrine pancreatic insufficiency (EPI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on presentation, genotype and/or sweat chloride
* Fecal elastase <100 mcg/g stool
* Good disease control with porcine PERT prior to enrollment
* Good nutritional status

Exclusion Criteria:

* History or diagnosis of fibrosing colonopathy
* Distal intestinal obstruction syndrome in 6 months prior to screening
* Receiving enteral tube feedings
* Chronic diarrheal illness unrelated to pancreatic insufficiency
* Liver abnormalities, or liver or lung transplant, or significant bowel resection
* Forced expiratory volume in 1 second (FEV1) <30%

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Coefficient of Fat Absorption (CFA) | 8 weeks
  Non-inferiority of Liprotamase to approved porcine PERT

SECONDARY OUTCOMES:
Coefficient of Nitrogen Absorption (CNA) | 8 weeks
  Non-inferiority of Liprotamase to approved porcine PERT
Safety, as measured by number of participants with adverse events or laboratory abnormalities | 6 months
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gangal, Study Director — Anthera Pharmaceuticals
Locations (50):
- United States (28):
  - Investigator Site 139, Little Rock, Arkansas
  - Investigator Site #123, Long Beach, California
  - Investigator Site 107, Los Angeles, California
  - Investigator Site 143, Orange, California
  - Investigator Site 150, Denver, Colorado
  - Investigator Site 147, Wilmington, Delaware
  - Investigator Site 117, Altamonte Springs, Florida
  - Investigator Site 102, Jacksonville, Florida
  - Investigator Site 130, Miami, Florida
  - Investigator Site 151, West Palm Beach, Florida
  - Investigator Site 110, Atlanta, Georgia
  - Investigator Site 109, Glenview, Illinois
  - Investigator Site 148, Iowa City, Iowa
  - Investigator Site #122, Louisville, Kentucky
  - Investigator Site 132, Portland, Maine
  - Investigator Site 124, Ann Arbor, Michigan
  - Investigator Site 140, Kalamazoo, Michigan
  - Investigator Site 134, Jackson, Mississippi
  - Investigator Site 135, Las Vegas, Nevada
  - Investigator Site 118, Durham, North Carolina
  - Investigator Site #103, Cleveland, Ohio
  - Site Investigator #113, Toledo, Ohio
  - Investigator Site 101, Oklahoma City, Oklahoma
  - Investigator Site 136, Oklahoma City, Oklahoma
  - Investigator Site 106, Hershey, Pennsylvania
  - Investigator Site 111, Dallas, Texas
  - Investigator Site 116, Houston, Texas
  - Investigator Site 112, Richmond, Virginia
- Hungary (4):
  - Investigator Site 302, Törökbálint, Pest County
  - Investigator Site 304, Mosdós, Somogy County
  - Investigator Site 306, Budapest
  - Investigator Site 307, Budapest
- Investigator Site 601, Jerusalem, Israel
- Lithuania (2):
  - Investigator Site 901, Kaunas
  - Investigator Site #902, Vilnius
- Poland (8):
  - Investigator Site 203, Karpacz
  - Site 206, Lodz
  - Investigator Site 201, Lublin
  - Investigator Site 205, Lublin
  - Investigator Site 202, Rabka-Zdrój
  - Investigator Site 209, Rzeszów
  - Investigator 204, Sopot
  - Investigator Site 210, Łomianki
- Spain (5):
  - Investigator Site 405, El Palmar, Murcia
  - Investigator Site 401, Madrid
  - Investigator Site 403, Madrid
  - Investigator Site 402, Málaga
  - Investigator Site 404, Valencia
- United Kingdom (2):
  - Investigatior Site 701, Southampton, Hampshire
  - Investigator Site 702, Exeter